CLINICAL TRIAL: NCT03573817
Title: A Phase 3b, 42-day, Randomized, Double-Blind, Placebo Controlled, Parallel Group Study to Evaluate the Safety and Tolerability of Nebulized Revefenacin and Nebulized Formoterol Fumarate (PERFOROMIST®) Administered in Sequence and as a Combined Solution in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: A 42-day Parallel Group Safety Study of Revefenacin and Formoterol, Administered in Sequence and as a Combination, in Participants With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0167
Record Dates: First submitted 2018-05-24; First posted 2018-06-29 (Actual); Results first posted 2019-12-18 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease; Pulmonary Function; COPD; Performist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — revefenacin; Formoterol Fumarate

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, parallel-group study. Each participant will receive treatment daily for a total of 42 days. One group will receive placebo and formoterol and one group will receive revefenacin and formoterol.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Period 1: Revefenacin + Formoterol (Sequential) (Experimental): Days 1 to 21: Revefenacin and formoterol will be sequentially administered in the morning. Formoterol will be administered again in the evening.
  Interventions: Drug: Revefenacin; Drug: Formoterol
- Period 2: Revefenacin + Formoterol (Combo Solution) (Experimental): Days 22 to 42: After a 21 day period, the participants from the Revefenacin + Formoterol (Sequential) Arm will be dosed for 21 days with a combination of revefenacin and formoterol administered as a combined solution. Formoterol will be administered again in the evening.
  Interventions: Drug: Revefenacin; Drug: Formoterol
- Period 1: Placebo + Formoterol (Sequential) (Placebo Comparator): Days 1 to 21: Placebo versions of revefenacin and formoterol will be sequentially administered in the morning. Formoterol will be administered again in the evening.
  Interventions: Drug: Placebo; Drug: Formoterol
- Period 2: Placebo + Formoterol (Combo Solution) (Placebo Comparator): Days 22 to 42: After a 21 day period, the participants from Placebo + Formoterol (Sequential) Arm the will be dosed for 21 days with a combination of placebo revefenacin and formoterol administered as a combined solution. Formoterol will be administered again in the evening.
  Interventions: Drug: Placebo; Drug: Formoterol

INTERVENTIONS:
Drug: Revefenacin — Revefenacin is administered via a nebulizer.
  Other Names: TD-4208
  Arms: Period 1: Revefenacin + Formoterol (Sequential); Period 2: Revefenacin + Formoterol (Combo Solution)
Drug: Placebo — Placebo version of Revefenacin is administered via a nebulizer.
  Arms: Period 1: Placebo + Formoterol (Sequential); Period 2: Placebo + Formoterol (Combo Solution)
Drug: Formoterol — Administered sequentially in both revefenacin and placebo arms using a nebulizer.

SUMMARY:
The primary objective of the study was to characterize the safety and tolerability of once-daily revefenacin inhalation solution when dosed sequentially with twice-daily formoterol inhalation solution (PERFOROMIST®) compared to PERFOROMIST®, in a population of participants with moderate-to-very severe Chronic Obstructive Pulmonary Disease (COPD) over 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a male or female subject 40 years of age or older.
* Participant is willing and able to provide signed and dated written informed consent.
* Participant has a current or past cigarette smoking history (or equivalent for cigar or pipe smoking history) of at least 10 pack-years.
* Participant must be willing and able to attend study visits according to the visit schedule and adhere to all study assessments/procedures.

Exclusion Criteria:

* Participant has a concurrent disease or condition that, in the opinion of the investigator, would interfere with study participation or confound the evaluation of safety, tolerability, or pharmacokinetics of the study drug.
* Participant has a history of reactions or hypersensitivity to inhaled or nebulized anticholinergics, short-acting beta-agonists and long-acting beta-agonists.
* Participant with clinically significant and uncontrolled hypertension, hypercholesterolemia or Type II diabetes mellitus, as assessed by the investigator.
* Participant is unwilling or unable to stop the use of prohibited medications during the washout (if required) and treatment period and follow-up period of the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (12):
- United States (12):
  - Theravance Biopharma Investigational Site, Miami, Florida
  - Theravance Biopharma Investigational Site, Orlando, Florida
  - Theravance Biopharma Investigational Site, Sarasota, Florida
  - Theravance Biopharma Investigational Site, Tampa, Florida
  - Theravance Biopharma Investigational Site, Saint Charles, Missouri
  - Theravance Biopharma Investigational Site, Monroe, North Carolina
  - Theravance Biopharma Investigational Site, Columbus, Ohio
  - Theravance Biopharma Investigational Site, Medford, Oregon
  - Theravance Biopharma Investigational Site, Erie, Pennsylvania
  - Theravance Biopharma Investigational Site, Gaffney, South Carolina
  - Theravance Biopharma Investigational Site, Greenville, South Carolina
  - Theravance Biopharma Investigational Site, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized 1:1 to one of two treatment groups and received treatment twice-daily for the two 21-day treatment periods. The participants in Arms 1 and 2 are the same (minus attrition), and the participants in Arms 3 and 4 are the same (minus attrition).
Groups:
- Revefenacin + Formoterol: Includes participants from Arm 1 (Day 1-21) and Arm 2 (Day 22-42).
- Placebo + Formoterol: Includes participants from Arm 3 (Day 1-21) and Arm 4 (Day 22-42).
Period: Overall Study
Arm/Group | Revefenacin + Formoterol | Placebo + Formoterol
Started | 63 | 59
Randomized and Treated With Study Drug | 63 | 59
Completed | 62 | 55
Not Completed | 1 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: 122 participants were enrolled in this study and received at least one dose of study drug. The disposition data is shown for the two different treatment types.
Groups:
- Total: Total of all reporting groups
Arm/Group | Revefenacin + Formoterol | Placebo + Formoterol | Total
Number analyzed (Participants) | 63 | 59 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (8.71) | 64.4 (8.43) | 63.7 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 35 | 34 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 56 | 56 | 112
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 60 | 56 | 116
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 63 | 59 | 122
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.22 (6.642) | 29.11 (6.349) | 29.17 (6.475)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced at Least One Treatment-Emergent Adverse Event
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a pharmaceutical product that did not necessarily have to have a causal relationship with this treatment. A treatment-emergent AE is an AE that occurred after the participant has received the study drug.
Time Frame: Day 1 to End of Period 2, a Maximum of 42 days + 7 days follow-up (Each period was 21 days)
Population: The populations for Arms 1 and 2 are made up of the same participants, however 4 participants dropped out prior to beginning Period 2. Similarly, the populations for Arms 3 and 4 are made up of the same participants, but one participant dropped out prior to beginning Period 2.
Measure: Count of Participants; unit: Participants
Groups:
- Period 1: Revefenacin + Formoterol (Sequential): Days 1 to 21: revefenacin and formoterol sequentially administered via nebulizer in the morning. Formoterol will be administered again in the evening.
  .
- Period 2: Revefenacin + Formoterol (Combo Solution): Days 22 to 42: After a 21 day period, the participants from the Revefenacin + Formoterol (Sequential) Arm will be dosed for 21 days with a combination of revefenacin and formoterol administered as a combined solution via a single nebulization. Formoterol will be administered again in the evening.
- Period 1: Placebo + Formoterol (Sequential): Days 1 to 21: Placebo versions of revefenacin and formoterol will be sequentially administered via nebulizer in the morning. Formoterol will be administered again in the evening.
- Period 2: Placebo + Formoterol (Combo Solution): Days 22 to 42: After a 21 day period, the participants from Placebo + Formoterol (Sequential) Arm the will be dosed for 21 days with a combination of placebo revefenacin and formoterol administered as a combined solution via a single nebulization. Formoterol will be administered again in the evening.
Arm/Group | Period 1: Revefenacin + Formoterol (Sequential) | Period 2: Revefenacin + Formoterol (Combo Solution) | Period 1: Placebo + Formoterol (Sequential) | Period 2: Placebo + Formoterol (Combo Solution)
Number analyzed (Participants) | 59 | 55 | 63 | 62
Participants | 7 | 6 | 3 | 5

2. Primary Outcome: Number of Participants Who Experienced at Least One Serious Treatment-Emergent Adverse Event
Description: A serious adverse event (SAE) was defined as any untoward medical occurrence occurring at any dose that resulted in any of the following outcomes:
  * Death
  * Life-threatening situation. "Life-threatening" refers to a situation in which the participant was at risk of death at the time of the event; it does not refer to an event which might have caused death if it were more severe
  * Inpatient hospitalization or prolongation of existing hospitalization
  * Congenital anomaly in the offspring of a participant who received study drug
  * Important medical events that may not result in death, be immediately life-threatening, or require hospitalization, could have been considered an SAE when, based upon appropriate medical judgment, they may have jeopardized the participant and may have required medical or surgical intervention to prevent one of the outcomes listed in this definition
  A treatment-emergent SAE is an SAE that occurred after the participant has received the study drug.
Time Frame: Day 1 to End of Period 2, a Maximum of 42 days + 7 days follow-up (Each period was 21 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Period 1: Revefenacin + Formoterol (Sequential): Days 1 to 21: Revefenacin and formoterol will be sequentially administered via nebulizer in the morning. Formoterol will be administered again in the evening.
Arm/Group | Period 1: Revefenacin + Formoterol (Sequential) | Period 2: Revefenacin + Formoterol (Combo Solution) | Period 1: Placebo + Formoterol (Sequential) | Period 2: Placebo + Formoterol (Combo Solution)
Number analyzed (Participants) | 59 | 55 | 63 | 62
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Relevant Changes in Vital Sign Measurements
Description: Clinically significant changes identified based on change from baseline. Vital signs measured included heart rate, systolic blood pressure and diastolic blood pressure.
Time Frame: Baseline to End of Period 2, a Maximum of 42 days + 7 days follow-up (Each period was 21 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Revefenacin + Formoterol (Sequential) | Period 2: Revefenacin + Formoterol (Combo Solution) | Period 1: Placebo + Formoterol (Sequential) | Period 2: Placebo + Formoterol (Combo Solution)
Number analyzed (Participants) | 59 | 55 | 63 | 62
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Relevant Changes in Clinical Laboratory Measurements
Description: Clinically relevant changes identified based on change from baseline. Laboratory Measures assessed included hematology and serum.
Time Frame: Baseline to End of Period 2, a Maximum of 42 days + 7 days follow-up (Each period was 21 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Revefenacin + Formoterol (Sequential) | Period 2: Revefenacin + Formoterol (Combo Solution) | Period 1: Placebo + Formoterol (Sequential) | Period 2: Placebo + Formoterol (Combo Solution)
Number analyzed (Participants) | 59 | 55 | 63 | 62
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Relevant Changes in Electrocardiogram Results
Description: Clinically relevant changes identified based on change from baseline.
Time Frame: Baseline to End of Period 2, a Maximum of 42 days + 7 days follow-up (Each period was 21 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Revefenacin + Formoterol (Sequential) | Period 2: Revefenacin + Formoterol (Combo Solution) | Period 1: Placebo + Formoterol (Sequential) | Period 2: Placebo + Formoterol (Combo Solution)
Number analyzed (Participants) | 59 | 55 | 63 | 62
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Period 1: Day 1 to Day 21; Period 2: Day 22 to 42 (+7 days follow-up)
Description: An adverse event was any untoward medical occurrence in a participant administered a pharmaceutical product that did not necessarily have to have a causal relationship with this treatment.
Arm/Group | Period 1: Revefenacin + Formoterol (Sequential) | Period 2: Revefenacin + Formoterol (Combo Solution) | Period 1: Placebo + Formoterol (Sequential) | Period 2: Placebo + Formoterol (Combo Solution)
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/55 | 0/63 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/55 | 0/63 | 0/62
Other Adverse Events (participants affected / at risk) | 3/63 | 5/62 | 7/59 | 6/55
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: Revefenacin + Formoterol (Sequential) (N=63) | Period 2: Revefenacin + Formoterol (Combo Solution) (N=62) | Period 1: Placebo + Formoterol (Sequential) (N=59) | Period 2: Placebo + Formoterol (Combo Solution) (N=55)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Sputum purulent (Infections and infestations) | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1
Muscle contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may communicate the trial results generated by the PI, but only after the first publication or presentation of the combined study results generated by all participating sites. The Sponsor can then review trial results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days. The Sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT03573817/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT03573817/SAP_001.pdf